CLINICAL TRIAL: NCT01913236
Title: A Pragmatic Cluster Randomised Trial of a Tailored Intervention for Implementing Recommendations for Managing Depressed Elderly Patients in Primary Care: Protocol
Brief Title: Tailored Implementation Intervention for Managing Depressed Elderly Patients in Primary Care
Acronym: TICD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sykehuset Innlandet HF (Other)
Collaborators: European Union (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 150204; 258837 (Other Grant/Funding Number: European Union Seventh Framework Program 2007-2013)
Record Dates: First submitted 2013-07-29; First posted 2013-08-01 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2013-07

CONDITIONS: Depression
Keywords: Tailored implementation interventions; Primary care; Depression in the elderly
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Implementation intervention (Experimental): Tailored implementation intervention to address determinants of practice in primary care
  Interventions: Other: Implementation intervention
- Control (No Intervention): Treatment as usual provided by general practitioners to elderly patients with depression

INTERVENTIONS:
Other: Implementation intervention — Investigators will provide a comprehensive package of interventions to assist health care professionals to adhere to the recommendations. The package will include support for developing a collaborative care plan in the municipality, resources for general practitioners and other health care professionals, resources for patients, their relatives and volunteers,outreach visits to general practitioners' practices and their educational groups, educational resources and web-based resources.
  Arms: Implementation intervention

SUMMARY:
Background The prevalence of depression is high and the elderly have an increased risk of developing a chronic course. International data suggest that depression in the elderly is under-recognised, the latency before clinicians provide a treatment plan is longer, and elderly patients with depression are not offered psychotherapy to the same degree as younger patients. Although recommendations for the treatment of elderly patients with depression exist, health care professionals adhere to these recommendations to a limited degree only. Investigators conducted a systematic review to identify recommendations for managing depression in the elderly and prioritised six recommendations. Investigators identified and prioritised determinants of practice related to implementation of these recommendations in primary care, and subsequently discussed and prioritised interventions to address the identified determinants. The objective of this study is to evaluate the effectiveness of these tailored implementation interventions to implement six recommendations for the management of elderly patients with depression in primary care.

Methods/design Investigators will conduct a pragmatic cluster randomised trial comparing implementation of the six recommendations using tailored interventions with usual care. Investigators will randomize 80 municipalities into one of two groups: an intervention group, to which investigators will deliver tailored interventions to implement the six recommendations, and a control group, to which investigators will not deliver any intervention. Investigators will randomise municipalities rather than patients, individual clinicians or practices because we will deliver the intervention for the first three recommendations at the municipal level and investigators want to minimise the risk of contamination across practices for the other three recommendations. The primary outcome is the proportion of general practitioners' behaviours which are consistent with the recommendations.

Discussion This trial will investigate whether a tailored implementation approach is an effective strategy to improve collaborative care in the municipalities and health care professionals' practice towards elderly patients with depression in primary care. The effectiveness evaluation described in this protocol will be accompanied with a process evaluation exploring why and how the interventions were effective or ineffective.

ELIGIBILITY:
Inclusion Criteria:

Home-dwelling patients aged 65 or higher, who have a diagnosis of depression, according to International Statistical Classification of Diseases and Related Health Problems, Tenth Revision

Exclusion Criteria:

Patients will be excluded if they have a diagnosis of dementia, bipolar disorder or reside in nursing homes or is assessed by their practitioner to have low life expectancy.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-09; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
General practitioners'adherence to treatment recommendations | 3-6 months after end of intervention

SECONDARY OUTCOMES:
Patient improvement | 3-6 months after end of intervention
  General practitioners' assessment of improvement
Patient improvement | 3-6 months after end of intervention
  Patients' assessment of improvement from depressive and anxiety symptoms, assessment of sleep, adherence to medication, physical exercise and problem-solving abilities

CONTACTS AND LOCATIONS:
Overall Officials: Michel Wensing, Professor, Principal Investigator
Locations (1):
- Knowledge Centre for the Health Services, Oslo, Oslo County, Norway

REFERENCES:
- [Background] Wensing M, Oxman A, Baker R, Godycki-Cwirko M, Flottorp S, Szecsenyi J, Grimshaw J, Eccles M. Tailored Implementation For Chronic Diseases (TICD): a project protocol. Implement Sci. 2011 Sep 7;6:103. doi: 10.1186/1748-5908-6-103. PMID 21899753
- [Background] Flottorp SA, Oxman AD, Krause J, Musila NR, Wensing M, Godycki-Cwirko M, Baker R, Eccles MP. A checklist for identifying determinants of practice: a systematic review and synthesis of frameworks and taxonomies of factors that prevent or enable improvements in healthcare professional practice. Implement Sci. 2013 Mar 23;8:35. doi: 10.1186/1748-5908-8-35. PMID 23522377
- [Background] Aakhus E, Flottorp SA, Oxman AD. Implementing evidence-based guidelines for managing depression in elderly patients: a Norwegian perspective. Epidemiol Psychiatr Sci. 2012 Sep;21(3):237-40. doi: 10.1017/S204579601200025X. Epub 2012 May 22. PMID 22793810
- [Background] Aakhus E, Granlund I, Odgaard-Jensen J, Oxman AD, Flottorp SA. A tailored intervention to implement guideline recommendations for elderly patients with depression in primary care: a pragmatic cluster randomised trial. Implement Sci. 2016 Mar 9;11:32. doi: 10.1186/s13012-016-0397-3. PMID 26956726
- [Background] Aakhus E, Granlund I, Oxman AD, Flottorp SA. Tailoring interventions to implement recommendations for the treatment of elderly patients with depression: a qualitative study. Int J Ment Health Syst. 2015 Sep 12;9:36. doi: 10.1186/s13033-015-0027-5. eCollection 2015. PMID 26366193
- [Background] Aakhus E, Oxman AD, Flottorp SA. Determinants of adherence to recommendations for depressed elderly patients in primary care: a multi-methods study. Scand J Prim Health Care. 2014 Dec;32(4):170-9. doi: 10.3109/02813432.2014.984961. Epub 2014 Nov 28. PMID 25431340
- [Derived] Aakhus E, Granlund I, Odgaard-Jensen J, Wensing M, Oxman AD, Flottorp SA. Tailored interventions to implement recommendations for elderly patients with depression in primary care: a study protocol for a pragmatic cluster randomised controlled trial. Trials. 2014 Jan 9;15:16. doi: 10.1186/1745-6215-15-16. PMID 24405891